CLINICAL TRIAL: NCT06264375
Title: E-SPORT: Evaluating the Sportive Potential Of Relevant New Talents - Development of a Specific Training Approach Based on Physical Activity for E-athletes and Gamers
Brief Title: Effect of a Specific and General Physical Exercise Intervention on Gaming and E-Sport Performance
Acronym: E-SPORT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E-SPORT
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Physical Activity
Keywords: e-sport; gaming; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 8 weeks of intervention, where Group 1 does a specific physical training, Group 2 a general physical training and Group 3 who does not train.
Masking Description: Data is collected and afterwards anonymized during the pre- and post measurement and during the intervention using a weekly questionnaire (activity level, gaming time)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Specific physical training (Experimental): 3 times training per week for approx. 30 minutes for 8 weeks. The training contains high intensity interval training (HIIT) elements. Moreover, exercises to improve grip strength, reaction times and anticipation are included.
  Interventions: Behavioral: Physical exercise
- General physical training (Experimental): 3 times training per week for approx. 30 minutes for 8 weeks. The training contains high intensity interval training (HIIT) elements.
  Interventions: Behavioral: Physical exercise
- No Training (No Intervention): Control group

INTERVENTIONS:
Behavioral: Physical exercise — see group description
  Arms: General physical training; Specific physical training

SUMMARY:
The goal of this randomized control intervention study is to test the effect of i) a specific physical training for e-sport and ii) a general physical training on e-sport performance, compared to iii) not training physically at all.

Participants are gamers and e-athletes who play at least >2hours peer week. The main questions it aims to answer are:

* Does physical training have an effect on e-sport related abilities (hand grip strength, reaction, anticipation)
* Does the training of specific elements, which aim at these abilities "out-game", transfer on the actual skills needed using a keyboard and mouse

Participants will be randomly - but mediated by hours of playing per week - distributed in 1 of 3 groups.

* Group 1 will 3 times per week for 30 minutes perform a specific physical training with focus on abilities needed in e-sport (grip strength, reaction, anticipation) over a timespan of 8 weeks.
* Group 2 will perform a similar physical training (load, intensity) to Group 1, but without specific elements.
* Group 3 will serve as control group without any training.

Researchers will compare Group 1, Group 2 and Groups 3 to see if the different trainings (Group 1 and Group 2) have different effect on e-sport performance and if no training (Group 3) differs in e-sport performance development.

DETAILED DESCRIPTION:
E-Sport is the competitive way of playing digital computer, console or smartphone games. Besides of this rational definition, it is a phenomenon which - not only because of the Covid-19 pandemic - received a lot of attention in the last couple of years. The high interest is often driven by the partially extraordinary high wages and price moneys offered to the involved actors, especially when compared to traditional sports. As an example, the 16 years old winner of the first Fortnite World Cup in 2019, Kyle "Bugha" Giersdorf, won 3 million dollar out of a 28.6 million dollar prize pool for succeeding in the final round. Besides of that, 19.000 people visited the event live in New York in the Arthur Ashe Stadium and 2.3 million watched it live via streams on YouTube and Twitch. Aside from the competitive e-sport environment, "gaming" can be described as the "hobby version", which has an even larger impact on an especially young generation. For example, in Austria 65% of the 18- to 64-year-old said in a survey in 2021 to play video-games on a weekly basis. Moreover, 25% stated to play at least 6 hours per week, some even more than 20 hours. When taking age into consideration, 2019 the share of gamers within the age group between 14 and 29 was 50%. Just like in other sports, casual and hobby gamers are influenced by elite (e-)sport athletes as role models. Hence, the behavior and especially the connection to physical activity of e-sport athletes can be particularly important, as it might have an influence on young e-sport or gaming affine individuals. Another fact is that the mentioned online streams become more and more the preferred media of the younger generations, turning their back on typical broadcast systems like TV or radio, what makes them hard to reach for e.g. public health advises broadcasted using the mentioned common channels. Besides the impressive numbers and the rapid growth of e-sport in recent years, there is a lack of research especially regarding the involvement of physical activity.

Regardless of the ongoing debate if e-sport should be considered as sport or not, research conducted about the effects of gaming on physical abilities could show that video-gaming supports hand-eye coordination, fine motor skills, enables e-athletes to perform up to 400 actions per minute using their keyboard and mouse, and enhances working memory performance and task-related cortical activity. Other research could show, that the level of performance in e-sport has a direct effect on the brain plasticity, presenting improved local functional integration within the executive areas of the brain of elite players compared to less-experienced e-athletes. Other arguments which support the idea of accepting e-sport as a sport, argue with mentioned elite eye-hand-coordination, fast reaction times in terms of visual information, and cognitive and strategic abilities over hours. Already in children, the visual abilities get trained by playing video-games as well, as research could show that spatial awareness could be improved by playing the game Tetris, or that movements of objects in a virtual space could be anticipated more efficiently. Other research about psychological factors and indicators in e-sport could show that attention, memory, information processing and task-switching are crucial parameters for e-sport athletes. All of this evidence proves that gaming affects the bodies and brains of an especially young population, as these are the major consumers of digital games on computers and consoles. Research about the effect of general physical activity on gaming performance presents that even a 6-minute rest including a non-sitting activity between games can have acute and chronic health benefits. Moreover, it improves processing speed and executive functions, which might beneficial for e-athletes during their games and competitions. With almost nine hours of physical activity per week, German e-athletes are considered as "active". Moreover, some e-athletes do train physically, however, not in a specific way and it remains topic to debate if this kind of training actually has an effect on their performance. Hence, the question arises if physical training towards skills and abilities, which are needed in e-sport, would be effective the other way around. Moreover, to investigate the effect of a general training of physical fitness could be of interest to 1) improve e-athletes' performance and 2) promote their health, as physical training would even more become a reasonable part of e-sport training. In more detail, research is missing regarding the question what specific physical and motor skills are needed in e-sport and if a specific training, which targets these abilities could be beneficial for e-athletes. To know about such possible synergy effects is necessary and of high interest, as 1) evidence-based information on this topic is scarce and 2) the number of e-athletes is increasing and measures should be taken to avoid injuries and promote performance and health in this community. As described already, e-sport is a phenomenon of the youth. Bringing physical activity in this community with the intention to help them improving their performance and preventing injuries, is an approach that urgently should be considered to ensure a healthier society in the future. One examples of potential synergies using physicality in e-sport is the hand grip strength, as there is evidence that a higher grip strength improves dexterity in elderly people. A better dexterity might be beneficial to perform game-specific actions with the fingers faster and more accurate, as needed in some game genres. A possible mechanism is the improved intramuscular coordination, which could be indicated by the higher force values and therefore be responsible for a better neuromuscular harmonization. The other way round, does video-gaming progress manual skills and grip strength of the non-dominant hand. Another example is the effect of gaming on cardiovascular and respiratory parameter like heart rate, respiratory rate and minute ventilation, which showed an increase during acute gaming. Interestingly the team with higher values performed better. The question arises, if the capability of withstanding higher heart rate thresholds or regenerating faster and coming "back to comfort" helps to increase performance in e-sport and gaming. That the energy expenditure during gaming is 40% higher than during sitting was shown already, stating that the physical fitness indeed has an impact on performance. However, if physical fitness has a measurable effect on gaming performance still needs to be evaluated. Other, especially coordinative abilities like reaction time are skills, which are often named first in the context of e-sport and gaming and have been shown to be similar for traditional sport athletes and e-athletes. Although there is a debate about the trainability of reaction, it appears that sport and e-sport do fasten reaction times. However, the possible effect of a training with focus on reaction time and its effect on e-sport and gaming performance still needs to be evaluated. In general there is evidence that e-sport and gaming are in need of specific motoric abilities, which are needed to succeed in certain games.

Results of the proposed project could be implemented in youth projects and schools and especially in physical education classes and an e-sport academy, which will be presented later. The great attention of young people regarding e-sport and gaming can be used as possibility to increase the awareness about living a healthy lifestyle. Hence, an evidence-based fundament is created to build up on. The implementation of physical activity in e-sports and gaming at an early state can be crucial to achieve a high acceptance in the community.

To conclude, the aim of the proposed project is to identify trainable parameters linked to physical activity, which are relevant in e-sport and gaming. The expected results are improvements in actual e-sport performance and e-sport related tasks achieved by a specific training. Moreover, it is expected to see an increase of performance due to a general training as well, compared to no physical training. Additionally, a specific physical training for e-athletes based on the obtained scientific evidence is to be developed. The resultant findings and advices can be used to promote the importance and advantages of physical activity in a young community, ultimately resulting in improved health awareness.

ELIGIBILITY:
Inclusion Criteria:

* playing video games on a regular basis (>2h per week)
* willing to take part in an 8 weeks intervention period containing physical training

Exclusion Criteria:

* any reasons which would make participation in physical activity impossible, such as acute injuries, chronic health problems or medical advices

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Grip Strength (Out-Game) | Baseline and week 8
  Grip strength of the hand measured in kg using the Takei Dynamometer 5401
Reaction Time (Out-Game) | Baseline and week 8
  Reaction time will be measured using a browser solution (aimbooster.com) and a 4-fold reaction test including 4 buttons which need to be pressed when a certain light shows up. Left upper corner light = left hand, right upper corner light = right hand, left lower corner light = left foot, right lower corner light = right foot. Per round, the lights will light up 10 times and the average reaction time will be calculated.
Anticipation (Out-Game) | Baseline and week 8
  The test is a horizontally moving laser, who differs in speed randomly. The test starts with ten left-to-right movements to get into the lasers' movement behavior, after which the actual test start. The task is to click on a button, just in the moment when the laser reaches the middle point, which is indicated by a "X" on the wall. The software detects the time difference for ten trials, if the click was performed too early, or too late respectively.
Whole Body Fitness | Baseline and week 8
  To test the ability of the participants to react not only using one movement, but combining different movements as a whole-body movement and fitness test, the BlazePods will be used. This training device consists of 4 so-called "pods", which are controlled by a smartphone application and enlighten in randomized order. The task is to tap upon the pod, as soon as it lights up. The test lasts 60 second, implementing a cardiovascular test.
Gaming Performance - Accuracy/Speed and Anticipation | Baseline and week 8
  Participants have to click on 1 of 3 visible circles which appear in the 3D surrounding of the game AimLab fpr 60 seconds. The task is to be as fast as possible in eliminating the circles, testing accuracy and speed of the participants. The AimLab software is a validated tool in measuring abilities needed in First-person-Shooters (FPS).
  A second task will be to track a circle which flicks randomly from one side to the other, again for 60 seconds. This ability is also needed in all FPS games.

SECONDARY OUTCOMES:
Well-being after training | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Participants of the experimental group are asked to rate their subjective wee-being on a 10-point likert scale before, during and after the exercise interventions

CONTACTS AND LOCATIONS:
Overall Officials: Felix Wachholz, PhD, Principal Investigator — Leopold-Franzens-Universität Innsbruck
Locations (1):
- Department of Sport Science, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Wachholz F, Gamper N, Schnitzer M. An 8-week physical exercise intervention for e'athletes improves physical performance rather than short-term esports performance parameters - a randomized controlled trial. Front Sports Act Living. 2025 Jan 21;6:1504205. doi: 10.3389/fspor.2024.1504205. eCollection 2024. PMID 39906318